CLINICAL TRIAL: NCT05996978
Title: Intensive Drug Therapy for Ischemic Stroke Caused by Severe Intracranial Arterial Stenosis
Status: Completed | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: No.2019-112
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive Drug Therapy: Dual antiplatelet therapy (DAPT) (aspirin 100 mg per day and clopidogrel 75 mg per day were administered for 90 days, followed by aspirin 100 mg per day for long term) and atorvastatin (40 mg per day for 14 days, followed by 20 mg per day long term) after enrollment.
  Interventions: Other: Intensive Drug Therapy

INTERVENTIONS:
Other: Intensive Drug Therapy — Observational only and no predesigned interventions in this study
  Other Names: observational only ,no intervention

SUMMARY:
To observe the safety and efficacy of intensive drug therapy for ischemic stroke caused by severe intracranial arterial stenosis.Patients with acute stroke caused by intracranial arterial stenosis (stenosis rate ≥70%) were enrolled and accept dual antiplatelet therapy (DAPT) (aspirin 100 mg/d and clopidogrel 75 mg/d for 90 days, followed by aspirin 100 mg/d for long term) under the guidance of platelet function analysis (Verifynow) combined with the intensive statin therapy (40 mg/d for 14 days, followed by 20 mg/d for long term).

DETAILED DESCRIPTION:
Patients (35 to 80 years ) with acute ischemic stroke, who can be treated within 72 hours of symptom onset will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomly selected.Patients were treated with dual antiplatelet therapy (DAPT) (aspirin 100 mg per day and clopidogrel 75 mg per day were administered for 90 days, followed by aspirin 100 mg per day for long term) and atorvastatin (40 mg per day for 14 days, followed by 20 mg per day long term) after enrollment. Patients with aspirin resistance (aspirin reaction units [ARU] ≥550) or clopidogrel resistance (P2Y12 reaction units [PRU] ≥208) were excluded on the 7th day of therapy.The primary objective is to observe the safety and efficacy of intensive drug therapy for ischemic stroke patients. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Ethics Committee of Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 80 years;
* Onset <72 hours;
* New-onset ischemic stroke confirmed by skull magnetic resonance diffusion weighted imaging (MR-DWI);
* Severe ICAS (stenosis ≥70%) indicated by time-of-flight magnetic resonance angiography (TOF-MRA).

Exclusion Criteria:

* Ischemic stroke caused by other etiological factors (e.g., cardio-embolism, arterial dissection, vasculitis, etc.);
* Post-infarction hemorrhagic transformation and intraplaque hemorrhage as indicated by imaging examination;
* Contraindications to aspirin, clopidogrel, or atorvastatin;
* Intracranial hemorrhage within 3 months and a recent history of surgery or trauma;
* Severe organ impairment, liver insufficiency, and renal insufficiency;
* Complicated with tumors or hemorrhagic diseases;
* Use of drugs forbidden to use in combination after onset, including other antiplatelet drugs, anticoagulants, thrombolytic drugs, and drugs affecting antiplatelet agents and statin metabolism.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute stroke caused by intracranial arterial stenosis (stenosis rate ≥70%)
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Characteristics of the vessel wall | 3 years
  The characteristics of the vessel wall were evaluated by high-resolution magnetic resonance imaging (HR-MRI).

SECONDARY OUTCOMES:
The change of the serum LDL-C level | 24 hours,14 days
  Low-density lipoprotein cholesterol (LDL-C) was tested in the laboratory before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Han, M.D., Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, China